CLINICAL TRIAL: NCT06001658
Title: Tumor Microenvironment Features of Response to Perioperative Gemcitabine, Cisplatin, and Pembrolizumab in Potentially Resectable Biliary Tract Cancers
Brief Title: Perioperative Gemcitabine, Cisplatin, and Pembrolizumab in Potentially Resectable Biliary Tract Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2390; IRB00371087 (Other: Johns Hopkins Medicine Internal Review Board)
Record Dates: First submitted 2023-08-08; First posted 2023-08-21 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Billiary Track Cancer
Keywords: Biliary Tract cancer; Pembrolizumab; Gemcitabine; Cisplatin; Immunotherapy; Potentially resectable biliary tract cancer; Anti PD-L1; PD-L1; Carcinoma
MeSH Terms: conditions — Biliary Tract Neoplasms; Carcinoma | interventions — Gemcitabine; Cisplatin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gemcitabine, Cisplatin and Pembrolizumab (Experimental)
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Gemcitabine — Patients will receive treatment on Day 1 and Day 8 of each cycle. Gemcitabine (1000 mg/m2) will be administered IV on Day 1 and Day 8 of each cycle, Q3 weeks with 2 - 4 cycles prior to surgery and then 4-6 cycles after surgery.
Drug: Cisplatin — Patients will receive treatment on Day 1 and Day 8 of each cycle. Cisplatin (25 mg/m2) will be administered IV on Day 1 and Day 8 of each cycle, Q3 weeks with 2 - 4 cycles prior to surgery and then 4-6 cycles after surgery.
Drug: Pembrolizumab — Patients will receive treatment on Day 1 of each cycle. Pembrolizumab (200 mg) will be administered IV on Day 1 of each cycle, Q3 weeks with 2 - 4 cycles prior to surgery and then 4-6 cycles after surgery. Pembrolizumab (400 mg) will be administered IV Q6 weeks up to 4 cycles as maintenance.
  Other Names: KEYTRUDA; anti-PD-1 mAb

SUMMARY:
The purpose of this study is to determine the safety of peri-operative gemcitabine, cisplatin, and pembrolizumab in patients with BTC, as well as whether the combination of gemcitabine, cisplatin, and pembrolizumab (gem/cis/pembro) is feasible and lead to pathologic responses.

ELIGIBILITY:
Inclusion Criteria:

* Must have a newly diagnosed, biopsy-proven biliary tract cancer (BTC) including gallbladder, intrahepatic, extrahepatic, and hilar cholangiocarcinoma.
* Resectable BTC (biliary tract cancer)
* Measurable disease per RECIST 1.1 as determined by the investigator.
* Age ≥18 years.
* ECOG (Eastern Cooperative Oncology Group) performance status ≤1 or Karnofsky ≥80
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests.
* Patients must have adequate liver function defined by study-specified laboratory tests.
* Patients with chronic or acute HBV or HCV infection must have disease controlled prior to enrollment.
* Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test.
* For both Women and Men, must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Receiving, or previously received, any systemic chemotherapy, or investigational agent for BTC.
* Has received prior radiotherapy within 2 weeks of start of study intervention.
* Patients with a history of prior treatment with anti-PD-1 and anti-PD-L1.
* Have been diagnosed with another cancer or myeloproliferative disorder whose natural history or treatment has the potential to interfere with safety or efficacy assessment of this study's investigational drugs.
* Has a known history of Human Immunodeficiency Virus (HIV)/AIDS
* Has active co-infection with HBV and HDV.
* Has a diagnosis of immunodeficiency.
* Has active autoimmune disease that has required systemic treatment in the past 2 years.
* Systemic or topical corticosteroids at immunosuppressive doses.
* Prior allogeneic stem cell transplantation or organ transplantation.
* Prior tissue or organ allograft or allogeneic bone marrow transplantation, including corneal transplants.
* Uncontrolled intercurrent active medical and/or psychiatric illness/social psychosocial problems that that would limit compliance with study requirements.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements.
* Evidence of clinical ascites.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Previously identified allergy or hypersensitivity to monoclonal antibodies or any component of the study treatment formulations.
* Pregnant or breastfeeding.
* WOCBP and men with female partners (WOCBP) who are not willing to use contraception.
* Subjects unable to undergo venipuncture and/or tolerate venous access.
* Patient is at the time of signing informed consent a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Average minimum Euclidean distance from CD8+ T cells to immunosuppressive tumor-associated macrophages (TAMs) at the per-cell level in patients with a major pathologic response versus pathologic non-responders. | 4 years
  The evaluable population of this endpoint consist of all patients who receive at least one dose of study drug and have TAMs and CD8 T cell measures at the time of surgery. TAMs being evaluated are the following: immunosuppressive TAMs with high Arginase-1 expression (CD68+CD163+Arg-1hiPDL1-/+), immunosuppressive TAMs with low Arginase-1 expression (CD68+CD163+Arg-1lo PDL1-/+), and less immunosuppressive TAMs (CD68+CD163-HLA-DRhi/CD86hi/PDL1hi)

SECONDARY OUTCOMES:
Number of participants experiencing grade 3 or above drug-related toxicities | 4 years
  When calculating the incidence of AEs, each AE (as defined by NCI CTCAE v5.0) will be counted only once for a given subject.
Number of patients proceeding to surgery without an extended treatment-related delay as a measure of feasibility | 144 days
  Extended treatment delay is defined as a delay of greater than 60 days of the pre-planned surgical evaluation date, or inability to go to surgery due to an adverse event related to study treatment.
Major pathologic response rate | 8-12 weeks
  The number of participants with a major pathologic response as defined by ≤ 10% residual viable tumor cells in the resection of the primary tumor and lymph nodes.
R0 resection rate | 60 days
  The number of participants with a R0 resection as defined by a microscopically margin-negative resection, in which no tumor (gross or microscopic) remains in the primary tumor bed.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Baretti, M.D., Principal Investigator — SKCCC Johns Hopkins Medical Institution
Locations (1):
- SKCCC Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No